CLINICAL TRIAL: NCT05595005
Title: Neural Bases of Post-stroke Emotion Perception Disorders
Acronym: STROKEM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_12; 2020-A00193-36 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Stroke Sequelae; Emotions
Keywords: stroke; emotions; neural bases
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke: Stroke patients (ischemic or hemorrhagic) in the chronic phase (> 6 months)
- Healthy controls: Healthy adult controls

SUMMARY:
This monocentric physiological study will evaluate the neural bases of visual recognition of emotions in stroke patients vs. healthy controls using MRI (functional and structural connectivity) and EEG.

DETAILED DESCRIPTION:
This monocentric physiological study will evaluate the neural bases of visual recognition of emotions in stroke patients vs healthy controls (2 groups of 40 subjects). It will include functional MRI, structural MRI (disconnectome), EEG, and behavioral assessments of emotion recognition and executive functions.

ELIGIBILITY:
Inclusion Criteria:

Stroke group:

* Man or Woman
* Age 18-80y
* Unique stroke, ischemic or hemorrhagic
* at the chronic phase (< 6 months)
* Written informed consent
* subject having a social insurance
* Subject who consent to complete all the study's experiments

Healthy controls group:

* Man or Woman
* Age 18-80y
* No history of neurological or psychiatric disease.

Exclusion Criteria:

Stroke group

* Subject who is unable to consent (due to dementia, severe aphasia, psychiatric disorder...)
* History of other neurologic disorders
* Significant le vel of depression or anxiety, assessed by the STAI and the BDI questionnaires
* Non corrected visual loss
* Subjects suffering from visual neglect (assessed by the Bells Test and a bisection test (20mm)
* contra-indications to MRI
* pregnant or breastfeeding woman
* Women of childbearing age without effective contraception

Healthy controls group

* Subject who is unable to consent (due to dementia, severe aphasia, psychiatric disorder...)
* History of neurologic disorders
* Significant level of depression or anxiety, assessed by the STAI and the BDI questionnaires
* Non-corrected visual loss
* contra-indications to MRI
* pregnant or breastfeeding woman
* Women of childbearing age without effective contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient group: 40 subjects Healthy control group: 40 subject
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
BOLD signal when fear visual recognition | 1 day
  Compare correlations of cerebral functional activations (BOLD) by fMRI between groups when stimulus = fear

SECONDARY OUTCOMES:
BOLD signal when happiness visual recognition | 1 day
  Compare correlations of cerebral functional activations (BOLD) by fMRI between groups when stimulus = happiness
Electrical connectivity (EEG) when fear visual recognition | 1 day
  Compare cerebral networks activated by a fear visual task recognition in both groups
Electrical connectivity (EEG) when fear happiness visual recognition | 1 day
  Compare cerebral networks activated by a happiness visual task recognition in both groups
Electrical connectivity (EEG) when emotions auditory recognition | 1 day
  Compare cerebral networks activated by an auditory task recognition in both groups
Relationship between behavioral performance and cerebral networks | 1 day
  Correlations between fMRI and EEG networks vs. behavioral performance (emotion recognition)
Structural connectivity | 1 day
  Disconnectome maps in the stroke patients group
Relationship between emotional self-assessment and cerebral networks | 1 day
  Correlation between the ESQ (emotional state questionnaire) and cerebral connectivity (EEG) and fMRI networks
Relationship between the behavioural performance in emotion recognition and executive functions | 1 day
  Correlation between behavioral performance in emotion recognition (Eckman Test) and executive functions (Stroop Test) in the stroke group
Relationship between lesion characteristics and the behavioral performance in emotion recognition | 1 day
  Correlation between lesion volume and the behavioural performance in emotion recognition (Eckman Test)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Allart, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Swynghedauw, Lille, France